CLINICAL TRIAL: NCT06411743
Title: A Phase II/III Clinical Study of Recombinant Human Albumin Injection for the Treatment of Hypoalbuminemia in Cirrhotic Patients With Ascites
Brief Title: Phase II/III of Recombinant Human Albumin Injection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ART-2021-005
Record Dates: First submitted 2024-03-29; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-03

CONDITIONS: Hepatic Ascites
Keywords: Hepatic Ascites
MeSH Terms: interventions — Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group1 (Experimental): Recombinant Human Albumin Injection,10g/day, once daily for 14 days
  Interventions: Biological: Recombinant Human Albumin Injection
- Treatment group2 (Experimental): Recombinant Human Albumin Injection,20g/day ,once daily for 7 days
  Interventions: Biological: Recombinant Human Albumin Injection
- Control group1 (Active Comparator): Human Albumin,10g/day, once daily for 14 days
  Interventions: Biological: Human Albumin
- Control group2 (Active Comparator): Human Albumin,20g/day, once daily for 7 days
  Interventions: Biological: Human Albumin

INTERVENTIONS:
Biological: Recombinant Human Albumin Injection — Recombinant Human Albumin injection, strength: 10 g/vial (20%, 50 mL); storage conditions: 2-8°C, protected from light; manufactured and supplied by Tonghua Anrate Biopharmaceutical Co., Ltd.
  Arms: Treatment group1; Treatment group2
Biological: Human Albumin — Human Albumin (An Pu Lai Shi®), strength: 10 g/vial (protein concentration 20%, 50 mL/vial), storage conditions: 2-8°C, protected from light; manufactured by Shanghai RAAS Blood Products Co., Ltd.
  Arms: Control group1; Control group2

SUMMARY:
This study was a Phase II/III multicenter, blinded, and positiveactive-controlled clinical study with seamless adaptive design to evaluate the dose-response relationship, safety, and immunogenicity of recombinant human albumin(rHA) injection for the treatment of hypoalbuminemia in cirrhotic patients with ascites, and to provide a reference for the design of the Phase III clinical study.

DETAILED DESCRIPTION:
This study was a Phase II/III multicenter, blinded, and positive-controlled clinical study with seamless adaptive design. The Phase II clinical study was conducted first, followed by the Phase III clinical study.The Phase II clinical study aimed to evaluate the dose-response relationship, safety, and immunogenicity of recombinant human albumin(rHA) injection for the treatment of hypoalbuminemia in cirrhotic patients with ascites, and provide a reference for the design of Phase III clinical study. Dosage: For the 10 g/day rHA injection group, the subjects were administered rHA at a dose of 10 g/day once daily for 14 days. For the 20 g/day rHA injection group, the subjects were administered rHA at a dose of 20 g/day once daily for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18-65 years (inclusive).
* Subjects with body weight ≥ 55.0 kg.
* Subjects who were diagnosed as liver cirrhosis with ascites according to the Guidelines for Diagnosis and Treatment of Liver Cirrhosis with Ascites and Related Complications (2017) issued by the Chinese Society of Hepatology CMA, with ascites graded 1-2 at diagnosis or after treatment, and also met the requirement of ALB < 30 g/L (based on test values on Day -14 to Day -3).
* Subjects who were able to understand and comply with the study procedures, voluntarily participated this study, and had signed the informed consent form (ICF).

Exclusion Criteria:

* Subjects with a history of allergies to biological products derived from Escherichia coli, yeast, or Chinese hamster ovary (CHO) cells, or blood products such as HSA.
* Subjects with hepatic encephalopathy of West-Haven HE Grade III or higher.
* Subjects with uncontrolled infections, such as body temperature > 37.5°C, white blood cell count > 9.5 × 10^9/L, or neutrophil percentage > 80% (including severe abdominal infection, upper respiratory tract infection, lower respiratory tract infection, urinary system infection, etc.).
* Subjects with a history of hepatorenal syndrome (HRS), or serum creatinine (Cr) > 2 × the upper limit of normal (ULN), or Cr increased by > 50% duringat screening period; or presence of urine protein 2+ or more.
* Subjects with other severe underlying conditions that, in the opinion of the investigator, affected the participation in this study, including but not limited to malignancies (except for liver cancer patients without portal vein or hepatic vein tumor thrombosis), complicated portal vein thrombosis, non-cirrhotic portal hypertension-related ascites, ischemic heart disease, stroke, chronic obstructive pulmonary disease, and Grade III-IV heart failure, and those with gastrointestinal bleeding who had stopped bleeding for less than 14 days after treatment or failed to stop bleeding after endoscopic variceal ligation.
* Subjects with organ transplant.
* Female subjects of childbearing potential who had a positive serum pregnancy test, or subjects refused to use contraceptive measures during the study.
* Subjects who had participated in other clinical trials and received investigational drugs within 3 months prior to screening.
* Subjects with abnormal laboratory test values:a.Hematology: platelets (PLT) < 30 × 10^9/L, hemoglobin (HGB) < 70 g/L;b.Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 5 × ULN, serum total bilirubin (TBIL) > 3 × ULN;c.Prothrombin activity < 40%, prothrombin time (PT) prolonged by > 5 seconds;d.Left ventricular ejection fraction (LVEF) < 50%.
* Subjects who were considered inappropriate for participation in the study by the investigator due to other reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in ALB | Day -1/7
  The change in ALB was determined by calculating the difference between the value measured after the last dose (immediately after the end of dosing) and the value measured before the first dose (the mean).

SECONDARY OUTCOMES:
Proportion of subjects with serum ALB level reaching 35 g/L at the end of administration | Day 7/14
  It referred to the proportion of subjects with serum ALB level ≥ 35 g/L at the end of dosing to the total number of subjects in that dose group.
Time taken to attain serum ALB of 35 g/L | Day1- Day7/14
  Defined as the time required from the first administration to serum ALB level ≥ 35 g/L.
Change from baseline in body weight of subjects at the end of administration | Day 7/14
  Change of body weight referred to the change in body weight after the end of dosing compared with the body weight on Day -1, which served as the baseline value. Please note that the body weight should be measured without urination under fasting conditions.
Change from baseline in abdominal circumference of subjects at the end of administration | Day 7/14
  It referred to the change in abdominal circumference at the end of treatment compared with the abdominal circumference on the last day of the pre-dose observation period, which served as a reference. Please note that the abdominal circumference should be measured without urination under fasting conditions.
Change from baseline in ascites depth of participantsubjects at the end of administration | Day 7/14
  It referred to the change in ascites depth at the end of dosing compared with the ascites depth on Day -1, which served as the baseline value.

CONTACTS AND LOCATIONS:
Overall Officials: Junqi Junqi, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University (Leading Site), Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No
The privacy of the participants will be kept strictly confidential to the investigator, the staff participating in the study, the sponsor, and the corresponding treatment. The study protocol, records, data, and all other information generated will be kept strictly confidential.